CLINICAL TRIAL: NCT01749007
Title: Assessment of Cognitive Functioning as it Relates to Risk for Suicide in Veterans With HIV/AIDS
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 12-1039
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2012-12

CONDITIONS: HIV/AIDS
Keywords: Veterans; HIV; AIDS; Cognitive Functioning; Suicide
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veterans with HIV/AIDS

SUMMARY:
The purpose of this project is to gather pilot data related to exploring relationships between cognitive impairment and/or psychiatric distress and suicidal thoughts and/or behaviors in Veterans with Human Immunodeficiency Virus (HIV)/Acquired Immune Deficiency Syndrome (AIDS). To achieve this goal, a neuropsychological battery will be administered to Veterans with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Veterans between ages 18 to 65
* Have a diagnosis of HIV/AIDS confirmed via medical record
* Currently receiving or eligible to receive physical and/or mental health care through the VA Eastern Colorado Health Care System

Exclusion Criteria:

* Acute intoxication via alcohol or other illicit drugs at time of assessment as determined by observation and/or interview.
* Psychosis at time of interview as determined by observation and/or interview.
* Poor Test of Memory Malingering (TOMM) performance (scores below 25 on Trial 1 or scores lower than 45 on Trial 2)
* Current status as a prisoner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans with HIV/AIDS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) | 1 Time Administration
  The WAIS-IV is a widely used and well established instrument used to assesses an individual's intellectual functioning within various cognitive domains and organizes performance into several indices including Verbal Comprehension Index, Perceptual Reasoning Index, Working Memory Index, and Processing Speed Index. A composite, Full Scale IQ, is also generated to represent an estimation of overall intellectual functioning.
Trail Making Test (TMT): Parts A & B | 1 Time Administration
  The TMT is a timed, pencil-paper, measure of attention, speed, and cognitive flexibility and requires participants to draw a line to accurately sequence 25 circles containing numbers (Part A) and alternating letters and numbers (Part B).
California Verbal Learning Test, Second Edition (CVLT-II) | 1 Time Adminstration
  The CVLT-II examines several aspects of verbal learning, organization, and memory.
Delis-Kaplan Executive Function System (D-KEFS) | 1 Time Administration
  Measure of executive functioning.
Brief VisuoSpatial Memory Test-Revised (BVMT-R) | 1 Time Administration
  The BVMT-R measures immediate and delayed visual memory.
Wisconsin Card Sorting Test (WCST) | 1 Time Administration
  Measure of executive functioning.
Outcome Questionnaire (OQ-45) | 1 Time Administration
  The OQ-45 is a 45-item questionnaire that was designed to measure key areas of mental health functioning (symptom distress, interpersonal functioning, and social role).
Beck Scale for Suicide Ideation (BSS) | 1 Time Administration
  The BSS is a 19-item scale that assesses severity of suicide ideation.

SECONDARY OUTCOMES:
Health Status Questionnaire (HSQ) | 1 Time Administration
  The HSQ is a 39-item, multiple choice, self-report measure that collects patient-reported, subjective data on eight subscales: Health Perception, Physical Functioning, Role Limitations/Physical Health, Role Limitations/Emotional Problems, Social Functioning, Mental Health, Bodily Pain and Energy/Fatigue.
University of Washington Risk Assessment Protocol-Revised (UWRAP) | 1 Time Administration
  The UWRAP will be used to address potential risk associated with participating in the study.
Test of Memory Malingering (TOMM) | 1 Time Administration
  The TOMM is a measure of effortful performance on objective tasks.
The Structured Clinical Interview for DSM-IV-Research Version (SCID-I) | 1 Time Administration
  The SCID is a reliable and valid semi-structured interview used to make psychiatric diagnosis in both clinical and research settings.
Lifetime Suicide Attempt Self Injury Interview (L-SASI) | 1 Time Administration
  The L-SASI was developed as a very brief survey of lifetime intentional self-harm behaviors and categorizes them into suicide attempts and non-suicidal acts.
Participant Demographics Form | 1 Time Administration
  A questionnaire was created by members of the research team to collect data regarding demographics.
Ohio State University TBI-ID (OSU TBI-ID) Short Form | 1 Time Administration
  The OSU TBI-ID Short Form will be used to determine history of TBI and presence of persistent TBI-related complaints.
Beck Hopelessness Scale (BHS) | 1 Time Administration
  The BHS is a 20-item true-false self-report scale that measures the level of negative expectations about the future held by respondents.
The Beck Depression Inventory (BDI-II) | 1 Time Administration
  The BDI-II is a widely used 21 item, self-administered instrument used to detect depression.
The Beck Anxiety Inventory (BAI) | 1 Time Administration
  The BAI is a widely-used, 21-item, self-administered instrument used to measure the severity of an individual's anxiety.
Military Suicide Research Consortium (MSRC) Common Data Elements | 1 Time Administration
  The Common Data Elements are a compilation of validated and reliable measures used to gather data on the risk factors for suicidal behavioral.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Signoracci, Ph.D., Principal Investigator — VISN 19 Denver VA MIRECC
Locations (1):
- Eastern Colorado Health Care System, Denver, Colorado, United States